CLINICAL TRIAL: NCT03609658
Title: Integrated Approach to Patient and Family Engagement for Advance Care Planning for Vulnerable Older Adult Within an Accountable Care Organization (ACO)
Brief Title: Integrated Multidisciplinary Patient and Family Advance Care Planning Trial
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00049370
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-06

CONDITIONS: Advance Care Planning
Keywords: Vulnerable Older Adults; Nurse Navigator; Usual Care; Family; Multimorbid patients

STUDY DESIGN:
Intervention Model Description: There are two groups. All participants are randomized prior to informed consent, and then only patients randomized to the interventional arm are approached for consent and subsequently enrolled in the intervention group. Note that patients that do not consent to the intervention are still counted as part of control group under an intent-to-treat paradigm, which necessitates passive ascertainment mechanisms for outcomes (i.e. administrative claims or the EHR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Navigator Pathway Group (Experimental): Participants in this Nurse Navigator led ACP pathway group will participate in ACP discussions, surveys, and participant visit(s) for duration of the study (12 months)
  Interventions: Behavioral: Nurse Navigator Pathway
- Usual Care Group (Sham Comparator): Participants in the Usual Care group will follow usual daily living activities for the duration of the study (12 months).
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Nurse Navigator Pathway — In the Nurse Navigator Pathway, nurse navigators are being used as leverage to: approach qualified patients to initiate advance care planning discussions, schedule advance care planning visit with patients' primary care provider to further discuss advance care planning and to mail advance care planning resources to patients after their initial advance care planning discussion.
  Arms: Nurse Navigator Pathway Group
Behavioral: Usual Care — In the Usual Care arm, there is no approach by nurse navigators to initiate advance care planning discussions and it does not have a structure advance care planning visit. Therefore, no further action is required for the patients who were randomly assigned to the usual care arm.
  Arms: Usual Care Group

SUMMARY:
The purpose of this study is to compare ways to engage sick patients and their family members in Advance Care Planning (ACP) discussions. Two pathways will be tested, discussions using a Nurse Navigator led pathway versus usual care.

DETAILED DESCRIPTION:
This study is a randomized, pragmatic, comparative effectiveness trial for determining better ways to engage multimorbid patients and their family members in Advance Care Planning through a Nurse Navigator led pathway versus usual care. Investigators propose to utilize Zelen's design (a more recent label/generalization for this type of design is the cohort multiple randomized controlled trial (cmRCT), a pragmatic clinical trial design whereby all participants are randomized prior to informed consent, and then only patients randomized to the interventional arm are approached for consent and subsequently enrolled in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or older patient within the Wake Forest/Cornerstone ACO
* Have seen their primary care provider within the Wake Forest/Cornerstone network in the past 12 months
* English speaking
* No documented Advance Directive in the EHR
* Impairments in either physical function, cognition, and/or frailty

Exclusion Criteria:

* No available proxy (e.g. in setting of cognitive impairment)
* Severe/advanced dementia
* Moderate to severe hearing loss
* Non-English speaking
* No phone number available for patient

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gabbard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (9):
- United States (9):
  - Family & Community Medicine of Asheboro, Asheboro, North Carolina
  - Claremont Family Medicine, Claremont, North Carolina
  - Conover Family Practice, Conover, North Carolina
  - Chronic Complex Care, High Point, North Carolina
  - Cornerstone Internal Medicine at Westchester, High Point, North Carolina
  - High Point Family Practice, High Point, North Carolina
  - Thomasville Family Practice, Thomasville, North Carolina
  - Downtown Health Plaza, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Census Bureau. International database. Table 094. Midyear population, by age and sex. Available at http://www.census.gov/population/www/projections/natdet-D1A.htmlExternal Web Site Icon.
- [Background] Gomez-Batiste X, Martinez-Munoz M, Blay C, Amblas J, Vila L, Costa X, Espaulella J, Espinosa J, Constante C, Mitchell GK. Prevalence and characteristics of patients with advanced chronic conditions in need of palliative care in the general population: a cross-sectional study. Palliat Med. 2014 Apr;28(4):302-11. doi: 10.1177/0269216313518266. Epub 2014 Jan 8. PMID 24403380
- [Background] "Methods for Analysis of the Financing and Use of Long-Term Services and Supports," supplemental material for Rising Demand for Long-Term Services and Supports for Elderly People (June 2013), www.cbo.gov/publication/44370.
- [Background] Schoenborn NL, Cayea D, McNabney M, Ray A, Boyd C. Prognosis communication with older patients with multimorbidity: Assessment after an educational intervention. Gerontol Geriatr Educ. 2017 Oct-Dec;38(4):471-481. doi: 10.1080/02701960.2015.1115983. Epub 2016 Feb 17. PMID 26885757
- [Background] Morrison RS. Research priorities in geriatric palliative care: an introduction to a new series. J Palliat Med. 2013 Jul;16(7):726-9. doi: 10.1089/jpm.2013.9499. Epub 2013 May 30. No abstract available. PMID 23721426
- [Background] Signorielli N: Physical disabilities, impairment and safety,mental illness, and death. In: Mass Media Images and Impact on Health: A Sourcebook. Westport, CT: Greenwood Press, 1993, pp. 37-42.
- [Background] Fortin M, Bravo G, Hudon C, Vanasse A, Lapointe L. Prevalence of multimorbidity among adults seen in family practice. Ann Fam Med. 2005 May-Jun;3(3):223-8. doi: 10.1370/afm.272. PMID 15928225
- [Background] Fortin M, Soubhi H, Hudon C, Bayliss EA, van den Akker M. Multimorbidity's many challenges. BMJ. 2007 May 19;334(7602):1016-7. doi: 10.1136/bmj.39201.463819.2C. PMID 17510108
- [Background] Marengoni A, Angleman S, Melis R, Mangialasche F, Karp A, Garmen A, Meinow B, Fratiglioni L. Aging with multimorbidity: a systematic review of the literature. Ageing Res Rev. 2011 Sep;10(4):430-9. doi: 10.1016/j.arr.2011.03.003. Epub 2011 Mar 23. PMID 21402176
- [Background] Smith SM, O'Dowd T. Chronic diseases: what happens when they come in multiples? Br J Gen Pract. 2007 Apr;57(537):268-70. No abstract available. PMID 17394728
- [Background] Taylor AW, Price K, Gill TK, Adams R, Pilkington R, Carrangis N, Shi Z, Wilson D. Multimorbidity - not just an older person's issue. Results from an Australian biomedical study. BMC Public Health. 2010 Nov 22;10:718. doi: 10.1186/1471-2458-10-718. PMID 21092218
- [Background] Vogeli C, Shields AE, Lee TA, Gibson TB, Marder WD, Weiss KB, Blumenthal D. Multiple chronic conditions: prevalence, health consequences, and implications for quality, care management, and costs. J Gen Intern Med. 2007 Dec;22 Suppl 3(Suppl 3):391-5. doi: 10.1007/s11606-007-0322-1. PMID 18026807
- [Background] Menotti A, Mulder I, Nissinen A, Giampaoli S, Feskens EJ, Kromhout D. Prevalence of morbidity and multimorbidity in elderly male populations and their impact on 10-year all-cause mortality: The FINE study (Finland, Italy, Netherlands, Elderly). J Clin Epidemiol. 2001 Jul;54(7):680-6. doi: 10.1016/s0895-4356(00)00368-1. PMID 11438408
- [Background] Fortin M, Lapointe L, Hudon C, Vanasse A, Ntetu AL, Maltais D. Multimorbidity and quality of life in primary care: a systematic review. Health Qual Life Outcomes. 2004 Sep 20;2:51. doi: 10.1186/1477-7525-2-51. PMID 15380021
- [Background] Townsend A, Hunt K, Wyke S. Managing multiple morbidity in mid-life: a qualitative study of attitudes to drug use. BMJ. 2003 Oct 11;327(7419):837. doi: 10.1136/bmj.327.7419.837. PMID 14551097
- [Background] Barnett K, Mercer SW, Norbury M, Watt G, Wyke S, Guthrie B. Epidemiology of multimorbidity and implications for health care, research, and medical education: a cross-sectional study. Lancet. 2012 Jul 7;380(9836):37-43. doi: 10.1016/S0140-6736(12)60240-2. Epub 2012 May 10. PMID 22579043
- [Background] Smith SM, Soubhi H, Fortin M, Hudon C, O'Dowd T. Managing patients with multimorbidity: systematic review of interventions in primary care and community settings. BMJ. 2012 Sep 3;345:e5205. doi: 10.1136/bmj.e5205. PMID 22945950
- [Background] Ryan A, Wallace E, O'Hara P, Smith SM. Multimorbidity and functional decline in community-dwelling adults: a systematic review. Health Qual Life Outcomes. 2015 Oct 15;13:168. doi: 10.1186/s12955-015-0355-9. PMID 26467295
- [Background] Iezzoni LI. Multiple chronic conditions and disabilities: implications for health services research and data demands. Health Serv Res. 2010 Oct;45(5 Pt 2):1523-40. doi: 10.1111/j.1475-6773.2010.01145.x. Epub 2010 Aug 2. PMID 21054370
- [Background] Quinones AR, Markwardt S, Botoseneanu A. Multimorbidity Combinations and Disability in Older Adults. J Gerontol A Biol Sci Med Sci. 2016 Jun;71(6):823-30. doi: 10.1093/gerona/glw035. Epub 2016 Mar 11. PMID 26968451
- [Background] Kogan AC, Wilber K, Mosqueda L. Person-Centered Care for Older Adults with Chronic Conditions and Functional Impairment: A Systematic Literature Review. J Am Geriatr Soc. 2016 Jan;64(1):e1-7. doi: 10.1111/jgs.13873. Epub 2015 Dec 2. PMID 26626408
- [Background] Connors MH, Sachdev PS, Kochan NA, Xu J, Draper B, Brodaty H. Cognition and mortality in older people: the Sydney Memory and Ageing Study. Age Ageing. 2015 Nov;44(6):1049-54. doi: 10.1093/ageing/afv139. PMID 26504121
- [Background] Bunn F, Goodman C, Burn AM. Multimorbidity and frailty in people with dementia. Nurs Stand. 2015 Sep 2;30(1):45-50. doi: 10.7748/ns.30.1.45.e9816. PMID 26329088
- [Background] Bunn F, Burn AM, Goodman C, Rait G, Norton S, Robinson L, Schoeman J, Brayne C. Comorbidity and dementia: a scoping review of the literature. BMC Med. 2014 Oct 31;12:192. doi: 10.1186/s12916-014-0192-4. PMID 25358236
- [Background] Campbell SE, Seymour DG, Primrose WR; ACMEPLUS Project. A systematic literature review of factors affecting outcome in older medical patients admitted to hospital. Age Ageing. 2004 Mar;33(2):110-5. doi: 10.1093/ageing/afh036. PMID 14960424
- [Background] Hagerty RG, Butow PN, Ellis PM, Lobb EA, Pendlebury SC, Leighl N, MacLeod C, Tattersall MH. Communicating with realism and hope: incurable cancer patients' views on the disclosure of prognosis. J Clin Oncol. 2005 Feb 20;23(6):1278-88. doi: 10.1200/JCO.2005.11.138. PMID 15718326
- [Background] Guiding principles for the care of older adults with multimorbidity: an approach for clinicians. Guiding principles for the care of older adults with multimorbidity: an approach for clinicians: American Geriatrics Society Expert Panel on the Care of Older Adults with Multimorbidity. J Am Geriatr Soc. 2012 Oct;60(10):E1-E25. doi: 10.1111/j.1532-5415.2012.04188.x. Epub 2012 Sep 19. No abstract available. PMID 22994865
- [Background] Herrin J, Harris KG, Kenward K, Hines S, Joshi MS, Frosch DL. Patient and family engagement: a survey of US hospital practices. BMJ Qual Saf. 2016 Mar;25(3):182-9. doi: 10.1136/bmjqs-2015-004006. Epub 2015 Jun 16. PMID 26082560
- [Background] Meghani SH, Hinds PS. Policy brief: the Institute of Medicine report Dying in America: Improving quality and honoring individual preferences near the end of life. Nurs Outlook. 2015 Jan-Feb;63(1):51-9. doi: 10.1016/j.outlook.2014.11.007. Epub 2014 Dec 11. PMID 25645482
- [Background] Zelen M. A new design for randomized clinical trials. N Engl J Med. 1979 May 31;300(22):1242-5. doi: 10.1056/NEJM197905313002203. PMID 431682
- [Background] Torgerson DJ, Roland M. What is Zelen's design? BMJ. 1998 Feb 21;316(7131):606. doi: 10.1136/bmj.316.7131.606. No abstract available. PMID 9518917
- [Background] Torgerson D. The use of Zelen's design in randomised trials. BJOG. 2004 Jan;111(1):2. doi: 10.1111/j.1471-0528.2004.00033.x. No abstract available. PMID 14687043
- [Background] House A, Knapp P. Informed consent. Trials that use Zelen's procedure should be acceptable. BMJ. 1997 Jul 26;315(7102):251. No abstract available. PMID 9253287
- [Background] Adamson J, Cockayne S, Puffer S, Torgerson DJ. Review of randomised trials using the post-randomised consent (Zelen's) design. Contemp Clin Trials. 2006 Aug;27(4):305-19. doi: 10.1016/j.cct.2005.11.003. Epub 2006 Feb 7. PMID 16455306
- [Background] Pate A, Candlish J, Sperrin M, Van Staa TP; GetReal Work Package 2. Cohort Multiple Randomised Controlled Trials (cmRCT) design: efficient but biased? A simulation study to evaluate the feasibility of the Cluster cmRCT design. BMC Med Res Methodol. 2016 Aug 26;16(1):109. doi: 10.1186/s12874-016-0208-1. PMID 27566594
- [Background] Rockwood K, Mitnitski A, Song X, Steen B, Skoog I. Long-term risks of death and institutionalization of elderly people in relation to deficit accumulation at age 70. J Am Geriatr Soc. 2006 Jun;54(6):975-9. doi: 10.1111/j.1532-5415.2006.00738.x. PMID 16776795
- [Background] Rockwood K, Mitnitski A. Frailty in relation to the accumulation of deficits. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):722-7. doi: 10.1093/gerona/62.7.722. PMID 17634318
- [Background] Pajewski NM, Williamson JD, Applegate WB, Berlowitz DR, Bolin LP, Chertow GM, Krousel-Wood MA, Lopez-Barrera N, Powell JR, Roumie CL, Still C, Sink KM, Tang R, Wright CB, Supiano MA; SPRINT Study Research Group. Characterizing Frailty Status in the Systolic Blood Pressure Intervention Trial. J Gerontol A Biol Sci Med Sci. 2016 May;71(5):649-55. doi: 10.1093/gerona/glv228. Epub 2016 Jan 11. PMID 26755682
- [Background] Drubbel I, de Wit NJ, Bleijenberg N, Eijkemans RJ, Schuurmans MJ, Numans ME. Prediction of adverse health outcomes in older people using a frailty index based on routine primary care data. J Gerontol A Biol Sci Med Sci. 2013 Mar;68(3):301-8. doi: 10.1093/gerona/gls161. Epub 2012 Jul 25. PMID 22843671
- [Background] Gonzalez-Colaco Harmand M, Meillon C, Bergua V, Tabue Teguo M, Dartigues JF, Avila-Funes JA, Amieva H. Comparing the predictive value of three definitions of frailty: Results from the Three-City study. Arch Gerontol Geriatr. 2017 Sep;72:153-163. doi: 10.1016/j.archger.2017.06.005. Epub 2017 Jun 17. PMID 28666213
- [Background] Rothman MD, Leo-Summers L, Gill TM. Prognostic significance of potential frailty criteria. J Am Geriatr Soc. 2008 Dec;56(12):2211-16. doi: 10.1111/j.1532-5415.2008.02008.x. PMID 19093920
- [Background] Roe L, Normand C, Wren MA, Browne J, O'Halloran AM. The impact of frailty on healthcare utilisation in Ireland: evidence from the Irish longitudinal study on ageing. BMC Geriatr. 2017 Sep 5;17(1):203. doi: 10.1186/s12877-017-0579-0. PMID 28874140
- [Background] Laniece I, Couturier P, Drame M, Gavazzi G, Lehman S, Jolly D, Voisin T, Lang PO, Jovenin N, Gauvain JB, Novella JL, Saint-Jean O, Blanchard F. Incidence and main factors associated with early unplanned hospital readmission among French medical inpatients aged 75 and over admitted through emergency units. Age Ageing. 2008 Jul;37(4):416-22. doi: 10.1093/ageing/afn093. Epub 2008 May 16. PMID 18487268
- [Background] Campitelli MA, Bronskill SE, Hogan DB, Diong C, Amuah JE, Gill S, Seitz D, Thavorn K, Wodchis WP, Maxwell CJ. The prevalence and health consequences of frailty in a population-based older home care cohort: a comparison of different measures. BMC Geriatr. 2016 Jul 7;16:133. doi: 10.1186/s12877-016-0309-z. PMID 27388294
- [Background] Gill TM, Allore HG, Gahbauer EA, Murphy TE. Change in disability after hospitalization or restricted activity in older persons. JAMA. 2010 Nov 3;304(17):1919-28. doi: 10.1001/jama.2010.1568. PMID 21045098
- [Background] Hubbard RE, Peel NM, Samanta M, Gray LC, Mitnitski A, Rockwood K. Frailty status at admission to hospital predicts multiple adverse outcomes. Age Ageing. 2017 Sep 1;46(5):801-806. doi: 10.1093/ageing/afx081. PMID 28531254
- [Background] Fried LP, Kronmal RA, Newman AB, Bild DE, Mittelmark MB, Polak JF, Robbins JA, Gardin JM. Risk factors for 5-year mortality in older adults: the Cardiovascular Health Study. JAMA. 1998 Feb 25;279(8):585-92. doi: 10.1001/jama.279.8.585. PMID 9486752
- [Background] Turner G, Clegg A; British Geriatrics Society; Age UK; Royal College of General Practioners. Best practice guidelines for the management of frailty: a British Geriatrics Society, Age UK and Royal College of General Practitioners report. Age Ageing. 2014 Nov;43(6):744-7. doi: 10.1093/ageing/afu138. PMID 25336440
- [Background] Bugarski V, Sakac V, Vodopivec S, Slankamenac P. Relation between personality dimensions and depressive symptoms in patients on hemodialysis. Med Pregl. 2010 May-Jun;63(5-6):305-12. doi: 10.2298/mpns1006305b. English, Serbian. PMID 21180270
- [Background] Clegg A, Bates C, Young J, Ryan R, Nichols L, Ann Teale E, Mohammed MA, Parry J, Marshall T. Development and validation of an electronic frailty index using routine primary care electronic health record data. Age Ageing. 2016 May;45(3):353-60. doi: 10.1093/ageing/afw039. Epub 2016 Mar 3. PMID 26944937
- [Background] Castanho TC, Amorim L, Zihl J, Palha JA, Sousa N, Santos NC. Telephone-based screening tools for mild cognitive impairment and dementia in aging studies: a review of validated instruments. Front Aging Neurosci. 2014 Feb 25;6:16. doi: 10.3389/fnagi.2014.00016. eCollection 2014. PMID 24611046
- [Background] Roccaforte WH, Burke WJ, Bayer BL, Wengel SP. Reliability and validity of the Short Portable Mental Status Questionnaire administered by telephone. J Geriatr Psychiatry Neurol. 1994 Jan-Mar;7(1):33-8. PMID 8192828
- [Background] Moorman SM, Carr D, Kirchhoff KT, Hammes BJ. An assessment of social diffusion in the Respecting Choices advance care planning program. Death Stud. 2012 Apr;36(4):301-22. doi: 10.1080/07481187.2011.584016. PMID 24567988
- [Background] Rietjens JA, Korfage IJ, Dunleavy L, Preston NJ, Jabbarian LJ, Christensen CA, de Brito M, Bulli F, Caswell G, Cerv B, van Delden J, Deliens L, Gorini G, Groenvold M, Houttekier D, Ingravallo F, Kars MC, Lunder U, Miccinesi G, Mimic A, Paci E, Payne S, Polinder S, Pollock K, Seymour J, Simonic A, Johnsen AT, Verkissen MN, de Vries E, Wilcock A, Zwakman M, van der Heide Pl A. Advance care planning--a multi-centre cluster randomised clinical trial: the research protocol of the ACTION study. BMC Cancer. 2016 Apr 8;16:264. doi: 10.1186/s12885-016-2298-x. PMID 27059593
- [Background] Yourman LC, Lee SJ, Schonberg MA, Widera EW, Smith AK. Prognostic indices for older adults: a systematic review. JAMA. 2012 Jan 11;307(2):182-92. doi: 10.1001/jama.2011.1966. PMID 22235089
- [Background] Sudore RL, Landefeld CS, Barnes DE, Lindquist K, Williams BA, Brody R, Schillinger D. An advance directive redesigned to meet the literacy level of most adults: a randomized trial. Patient Educ Couns. 2007 Dec;69(1-3):165-95. doi: 10.1016/j.pec.2007.08.015. Epub 2007 Oct 17. PMID 17942272
- [Background] Sudore RL, Barnes DE, Le GM, Ramos R, Osua SJ, Richardson SA, Boscardin J, Schillinger D. Improving advance care planning for English-speaking and Spanish-speaking older adults: study protocol for the PREPARE randomised controlled trial. BMJ Open. 2016 Jul 11;6(7):e011705. doi: 10.1136/bmjopen-2016-011705. PMID 27401363
- [Background] http://www.gotplans123.org/.
- [Background] Ito M, Nakajima S, Fujisawa D, Miyashita M, Kim Y, Shear MK, Ghesquiere A, Wall MM. Brief measure for screening complicated grief: reliability and discriminant validity. PLoS One. 2012;7(2):e31209. doi: 10.1371/journal.pone.0031209. Epub 2012 Feb 14. PMID 22348057
- [Background] Shear KM, Jackson CT, Essock SM, Donahue SA, Felton CJ. Screening for complicated grief among Project Liberty service recipients 18 months after September 11, 2001. Psychiatr Serv. 2006 Sep;57(9):1291-7. doi: 10.1176/ps.2006.57.9.1291. PMID 16968758
- [Background] Mori M, Yoshida S, Shiozaki M, et al.
- [Background] Yamaguchi T, Maeda I, Hatano Y, Mori M, Shima Y, Tsuneto S, Kizawa Y, Morita T, Yamaguchi T, Aoyama M, Miyashita M. Effects of End-of-Life Discussions on the Mental Health of Bereaved Family Members and Quality of Patient Death and Care. J Pain Symptom Manage. 2017 Jul;54(1):17-26.e1. doi: 10.1016/j.jpainsymman.2017.03.008. Epub 2017 Apr 24. PMID 28450216
- [Background] Glidden DV, Vittinghoff E. Modelling clustered survival data from multicentre clinical trials. Stat Med. 2004 Feb 15;23(3):369-88. doi: 10.1002/sim.1599. PMID 14748034
- [Background] Fine, J., & Gray, R. (1999). A Proportional Hazards Model for the Subdistribution of a Competing Risk. Journal of the American Statistical Association, 94(446), 496-509. doi:10.2307/2670170.
- [Background] Dong H, Robison LL, Leisenring WM, Martin LJ, Armstrong GT, Yasui Y. Estimating the burden of recurrent events in the presence of competing risks: the method of mean cumulative count. Am J Epidemiol. 2015 Apr 1;181(7):532-40. doi: 10.1093/aje/kwu289. Epub 2015 Feb 17. PMID 25693770
- [Background] Prentice R, Williams B, and Peterson A. On the regression analysis of multivariate failure time data. Biometrika 1981;68:373-379. .
- [Background] Julious SA. Sample Sizes for Clinical Trials. Chapman & Hall/CRC, Boca Raton, FL, 2010.
- [Background] Reeves D, Howells K, Sidaway M, Blakemore A, Hann M, Panagioti M, Bower P. The cohort multiple randomized controlled trial design was found to be highly susceptible to low statistical power and internal validity biases. J Clin Epidemiol. 2018 Mar;95:111-119. doi: 10.1016/j.jclinepi.2017.12.008. Epub 2017 Dec 19. PMID 29277558
- [Background] Sudore RL, Boscardin J, Feuz MA, McMahan RD, Katen MT, Barnes DE. Effect of the PREPARE Website vs an Easy-to-Read Advance Directive on Advance Care Planning Documentation and Engagement Among Veterans: A Randomized Clinical Trial. JAMA Intern Med. 2017 Aug 1;177(8):1102-1109. doi: 10.1001/jamainternmed.2017.1607. PMID 28520838
- [Derived] Gabbard J, Pajewski NM, Callahan KE, Dharod A, Foley KL, Ferris K, Moses A, Willard J, Williamson JD. Effectiveness of a Nurse-Led Multidisciplinary Intervention vs Usual Care on Advance Care Planning for Vulnerable Older Adults in an Accountable Care Organization: A Randomized Clinical Trial. JAMA Intern Med. 2021 Mar 1;181(3):361-369. doi: 10.1001/jamainternmed.2020.5950. PMID 33427851
- [Derived] Gabbard J, Pajewski NM, Callahan KE, Dharod A, Foley K, Ferris K, Moses A, Grey C, Williamson J. Advance care planning for vulnerable older adults within an Accountable Care Organization: study protocol for the IMPACT randomised controlled trial. BMJ Open. 2019 Dec 15;9(12):e032732. doi: 10.1136/bmjopen-2019-032732. PMID 31843844

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This protocol has Zelen's Design. Subjects were randomized to either the usual care arm or the nurse navigator arm prior to signing consent. And only those who were randomized to nurse navigator arm were consented. 379 subjects randomized to the nurse navigator arm, and of those, only 146 agreed to participate and signed consent. Subjects randomized to the usual care arm had a waiver of consent. The study team only did chart analysis for usual care subjects.
Period: Overall Study
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group
Started | 379 | 380
Completed | 379 | 380
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes all randomized subjects prior to signing consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group | Total
Number analyzed (Participants) | 379 | 380 | 759
Age, Customized [Count of Participants; unit: Participants]
  65 to <75 years | 149 | 156 | 305
  75 to <85 years | 161 | 151 | 312
  ≥85 years | 69 | 73 | 142
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 229 | 455
  Male | 153 | 151 | 304
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 300 | 317 | 617
  black | 71 | 59 | 130
  other | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 379 | 380 | 759

OUTCOME MEASURES:

1. Primary Outcome: Number of Patient's Documented Advance Care Planning Discussion- Nurse Navigator
Description: Reported as the number of documentations completed in the newly created ACP note template for nurse navigator note templates.
Time Frame: End of Study (Month 13)
Population: This outcome includes all randomized subjects (Zelen's design).
Measure: Number; unit: Discussions
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group
Number analyzed (Participants) | 379 | 380
Discussions | 134 | 0

2. Primary Outcome: Number of Patient's Documented Advance Care Planning Discussions - Provider
Description: Reported as the number of documentations completed in the newly created ACP note template for provider note templates.
Time Frame: End of Study (Month 13)
Population: This outcome applies to randomized subjects.
Measure: Number; unit: discussions
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group
Number analyzed (Participants) | 379 | 380
discussions | 160 | 14

3. Primary Outcome: Quality of Advance Care Planning Discussion - Nurse Navigator
Description: Measured by the newly created ACP note template for both nurse navigator (score ranging from 0-8). Score of 5 or higher determines better outcome.
Time Frame: End of Study (Month 13)
Population: Data was not collected for this outcome measure.
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Quality of Advance Care Planning Discussion - Provider
Description: Measured by the newly created ACP note template for provider note templates (score ranging from 0-15). Score of 8 or higher in the provider template determines better outcome.
Time Frame: End of Study (Month 13)
Population: data was not collected for this outcome
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Quality of Advance Care Planning Discussion From the Patient's Perspective
Description: Measured by the Quality about End of Life (EOL) Communication (QOC), The instrument is reported as 2 subscales: "general communication skills" and "communication about end-of-life care." Score range for the subscales is 1-11 Higher scores determine better outcomes.
Time Frame: End of Study (Month 13)
Population: This outcome does not apply to usual care group. Ten subjects were lost to follow up and 5 subjects withdrew consent from Nurse Navigator arm. Completion of the QOC was optional for the participants who had completed the provider visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group
Number analyzed (Participants) | 87 | 0
score on a scale
  General Communication | 10.2 (1.8) |
  End of Life | 7.9 (3.1) |

6. Secondary Outcome: Advance Care Planning Billing Code Usage
Description: ACP billing codes: 99497 and 99498 usages will be recorded
Time Frame: End of Study (Month 13)
Population: This outcome uses all randomized subjects (Zelen's Design).
Measure: Number; unit: code usages
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group
Number analyzed (Participants) | 379 | 380
code usages | 96 | 5

7. Secondary Outcome: Number of Designated Surrogate Decision Makers
Description: Reported as the number of designated surrogate decision makers documented in Electronic Health Record (EHR).
Time Frame: End of Study (Month 13)
Population: This outcome uses all randomized (Zelen's Design).
Measure: Number; unit: surrogate decision makers
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group
Number analyzed (Participants) | 379 | 380
surrogate decision makers | 241 | 132

8. Secondary Outcome: Advance Directive Completion
Description: Reported as the number of scanned advance directive documents in the EHR.
Time Frame: End of Study (Month 13)
Population: Based on all randomized (Zelen's Design).
Measure: Number; unit: scanned documents
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group
Number analyzed (Participants) | 379 | 380
scanned documents | 92 | 38

9. Other Pre Specified Outcome: Number of Medical Scope of Treatment (MOST) Discussions
Description: Reported as the number of completed MOST discussion within the new ACP template and/or scanned form in the EHR
Time Frame: End of Study (Month 13)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: After-death Bereaved Family Member Interview
Description: The After-death bereaved family member interview measures the quality of end of life care. Interview is analyzed utilizing Q-pro software for qualitative data.
Time Frame: Month 29
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Frequency of Patient Healthcare Utilization
Description: Frequency is measured by the number of healthcare events recorded in the EHR.
Time Frame: End of Study (Month 13)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Cost of Patient Healthcare Utilization
Description: Cost of patient healthcare utilization per group
Time Frame: End of Study (Month 13)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Provider Satisfaction With the Intervention Scale
Description: This is a likert scale total score (0-78). Higher scores denotes better outcomes
Time Frame: Month 11
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Number of Protocol Deviations
Description: The number of protocol deviations will be reported to measure the fidelity of study implementation.
Time Frame: End of Study (Month 13)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Usability of the ACP Documentation Tool (ACPWiseTool)
Description: Measured by the System Usability Scale (SUS) survey. Likert Scale of strongly disagree, disagree, neutral, agree, and strongly agree. Score ranges from 1 to 5. Higher score equates higher usability.
Time Frame: End of Study (Month 13)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Month 1 through Month 12
Description: Usual Care Group did not sign consent. No Adverse Events (AEs)/Serious Adverse Events (SAEs)/All-Cause Mortality data was collected for that arm.
Arm/Group | Nurse Navigator Pathway Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/379 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/379 | 0/0
Other Adverse Events (participants affected / at risk) | 0/379 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT03609658/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT03609658/ICF_001.pdf